CLINICAL TRIAL: NCT06821568
Title: Long-term Home-based Transcranial Electrical Stimulation for Cognitive and Motor Function in Older Adults With an Increased Risk of Dementia: a Randomized Controlled Trial
Brief Title: Home-Based Brain Stimulation for Motoric Cognitive Risk Syndrome
Acronym: TDCS4MCR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, Brad Manor, Associate Scientist, Hebrew SeniorLife
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00072642; 1R01AG081349-01A1 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-02-12 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease and Related Dementias; Cognition; Mobility Disability
Keywords: Anatomy; Anxiety; Atrophic; Behavioral; Brain; Brain Region; Cephalic; Cognitive; Communities; Dementia; Development; Dose; Double-Blind Method; Electric Stimulation; Enrollment; Evaluation; Exhibits; Exposure to; Frequencies; Future; Gait; Gait Speed; Genetic Crossing Over; Home; Impaired Cognition; Individual; Intervention; Intervention Studies; Magnetic Resonance Imaging; Measurable; Measures; Mood; Motor; Multi-Institutional Clinical Trial; Neuronal Plasticity; Outcome; Participant; Performance; Phase; Pilot Projects; Prefrontal Cortex; Randomized; Randomized Controlled Clinical Trials; Research; Resolution; Rest; Risk; Series; Site; Structure; Testing; Therapeutic; Time; Syndrome; Walking; Work; Arm; cerebral atrophy; Clinically relevant; cognitive task; Cost; Dementia Risk; Design; Executive Function; functional improvement; functional near infrared spectroscopy; Gray Matter; high risk; home test; improved; insight; late life; mental function; neural network; neuroimaging; noninvasive brain stimulation; normal aging; older adult; older men; older women; open label; primary endpoint; response; secondary outcome; smartphone application; transcranial direct current stimulation; trial design; walking speed; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Anxiety Disorders; Atrophy; Behavior; Dementia; Cognition Disorders; Syndrome

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a multi-site, sham-controlled, double-blinded, randomized trial of home-based tDCS with stimulation parameters tailored to target the anatomically defined left dlPFC of each participant. Participants will complete baseline cognitive and physical functioning assessments, as well as a structural MRI of the brain. After an initial open-label 2-week tDCS intervention, participants will be randomized into a tDCS arm (5 weekly tDCS sessions for 6 months), or a combination arm of 5 weekly tDCS sessions for 3 months before or after 5 weekly sessions of sham for 3 months via permuted block randomization stratified by sex to ensure that equal number of men and women are randomized to each intervention arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study personnel administering assessments, caregivers administering tDCS and the participants will not be aware of tDCS intervention arm assignment. The investigators will ensure double-blinding by programming the tDCS software with intervention-specific stimulation codes, as supplied by personnel uninvolved in data collection prior to study initiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalized Transcranial Direct Current Stimulation (tDCS) (Experimental): After an initial open-label 2-week home-based transcranial direct current stimulation (tDCS) intervention, participants will receive 5 weekly home-based tDCS sessions for 6 months. Baseline MRIs will enable personalization of tDCS via current flow modeling for optimization to each participant with the goal of generating an average electric field of 0.25 V/m within their identified left dlPFC. The direct current delivered by any one electrode will not exceed 2.0 mA and the total amount of current from all electrodes will not exceed 4 mA. Each 20-minute session will begin and end with a 60-second ramp up/down of current amplitude to maximize comfort.
  Interventions: Other: Personalized Transcranial Direct Current Stimulation (tDCS)
- Combination Arm; Sham Plus Personalized Transcranial Direct Current Stimulation (tDCS) (Active Comparator): After an initial open-label 2-week home-based transcranial direct current stimulation (tDCS) intervention, participants will receive a combination arm of five weekly tDCS sessions for 3 months before or after five weekly sessions of sham for 3 months. The investigators will use an active sham in which very low-level currents (0.5 mA total) will be transferred between electrodes in close proximity on the scalp throughout the entire 20-minute session. This intervention will be optimized to each participant to deliver currents designed to not significantly influence their cortical tissue, but still mimic the cutaneous sensations induced by tDCS. Participants in the combination arm will not know whether they are receiving tDCS or sham during the first or second 3-month period.
  Interventions: Other: Personalized Transcranial Direct Current Stimulation (tDCS); Other: Active-Sham

INTERVENTIONS:
Other: Personalized Transcranial Direct Current Stimulation (tDCS) — Home-based transcranial direct current stimulation (tDCS) tailored to target the left dlPFC.
Other: Active-Sham — Stimulation administered in very low-level currents (0.5 mA total) designed to not significantly influence cortical tissue, but still mimic the cutaneous sensations induced by tDCS.
  Arms: Combination Arm; Sham Plus Personalized Transcranial Direct Current Stimulation (tDCS)

SUMMARY:
The objective of this study is to determine the effects of a 6-month, home-based personalized transcranial direct current stimulation (tDCS) intervention targeting the left dorsolateral prefrontal cortex on cognitive function, dual task standing and walking, and other metrics of mobility in older adults with motoric cognitive risk syndrome (MCR).

DETAILED DESCRIPTION:
In older adults, motoric cognitive risk (MCR) is a pre-dementia transition state between "normal" aging and dementia. MCR is associated with impaired function within several brain networks that causes numerous symptoms including loss of memory, the ability to complete complex mental tasks, and the capacity to control one's walking and thus avoid falling and fall-related injuries. This study seeks to assess the short-term and long-term use of an investigational device called a transcranial direct current stimulation (tDCS).

tDCS is a noninvasive technology that enables selective modulation of brain network function, to provide multi-symptom relief to older adults with MCR. By using state-of-the-art technology to 1) utilize a personalized tDCS intervention via an established optimization approach using individual brain MRIs, and 2) complete stimulation in a home-based setting, this study is expected to result in the development of tDCS interventions that have maximal impact on daily life function within this population.

In this study, investigators will conduct a 9-month sham-controlled, double-blinded, multi-site trial in 128 older adults aged 65-90 years old with MCR. All enrolled participants will complete an open-label 2-week, 10-session tDCS intervention. During the open-label phase of the study, all participants will receive active tDCS. Then, participants will be randomly assigned into either the tDCS arm that receives five weekly tDCS sessions for 6 months, or a combination arm of five weekly tDCS sessions for 3 months before or after five weekly sessions of sham for 3 months. Sham treatment is similar to the study tDCS treatment, but omits the key therapeutic element of the treatment being studied. Participants in the combination arm will not know whether they are receiving tDCS or sham during the first or second 3-month period. Enrolled participants will complete assessments relating to cognition, mood, balance, and memory at baseline, after the 2-week open-label phase, after 3 and 6 months of tDCS, and again 3 months later. Once a week, participants will also complete a gait (walking) assessment at home. MRI scans will be performed at baseline and after completing 3 months of tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 65-90 years
* Subjective cognitive complaints as defined by a 'Yes' response to "Do you feel that you have more problems with memory than most?" or a 'No' response to "is your mind as clear as it used to be?"
* Montreal Cognitive Assessment (MoCA) score ≥21
* Slow gait speed as measured by averaging two 4-Meter walks and defined as a usual walking speed one standard deviation below age and sex-adjusted means.
* Absence of significant disability as defined by the ability to walk over the instrumented gait mat unassisted (e.g., able to walk without any walking aids for at least 2 minutes non-stop) and preserved activities of daily living as defined by a score of less than 9 on the Functional Activities Questionnaire.
* Identification of an eligible informant
* Identification of a willing and able tDCS-administrator; i.e., a study partner to lead the administration of home-based transcranial direct current stimulation (tDCS)
* Access to reliable WiFi in the participant's home

Exclusion Criteria:

* Formal education less than the 8th grade
* Previous physician diagnosis of dementia
* Any current diagnosis of a major psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depressive disorder)
* Evidence of moderate-to-severe depressive symptoms defined by a score of ≥9 on the 15-item Geriatric Depression Scale
* History of head trauma resulting in prolonged loss of consciousness
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, or immediate (first-degree relative) family history of epilepsy except for a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Hospitalization within the past three months due to acute illness, or as the result of a musculoskeletal injury significantly affecting gait or balance
* Any unstable medical condition or chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.) or study complication
* Substance use disorders within the past six months
* A hairstyle or headdress that prevents electrode contact with the scalp or would interfere with the stimulation (for example thick braids, hair weave, afro, wig)
* Chronic vertigo
* Myocardial infarction within the past 6 months
* Active cancer for which chemo-/radiation therapy is being received
* Legal blindness
* Visual hallucinations (history or self-report)
* Pacemaker
* Contraindications to MRI or tDCS, including unprovoked seizure within the past two years, risk of ferromagnetic objects anywhere in the body, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemaker, etc.), the presence of any active dermatological condition, such as eczema, on the scalp, etc. as outlined by current recommendations for noninvasive brain stimulation endorsed by the International Federation for Clinical Neurophysiology.
* History of REM sleep behavior disorder (RBD), often an early sign of Parkinson's disease
* Medications and medical history will be reviewed by the responsible covering physician and a decision about inclusion will be made based on the participant's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other CNS active drugs.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Dual task cost to gait speed | Pre-randomization baseline; within three days of completing the initial open-label tDCS intervention; Month 3, Month 6; Month 9.
  This metric assesses the degree to which performing a secondary cognitive task diminishes the control of gait.

SECONDARY OUTCOMES:
Executive function composite score | Baseline, within three days of completing initial open-label tDCS intervention, Month 3, Month 6, & Month 9.
  This metric is derived from the CANTAB computerized test battery and reflects age-, sex-, and education-based z-scores on numerous cognitive functions associated with executive function.
Dual task gait speed | Baseline, within three days of completing initial open-label tDCS intervention, Month 3, Month 6, & Month 9.
  This metric assesses the ability to walk and perform a cognitive task at the same time and predicts cognitive decline and the development of dementia.
Preferred gait speed | Baseline, within three days of completing initial open-label tDCS intervention, Month 3, Month 6, & Month 9.
  This metric assesses the preferred gait speed over the course of 4 meters.
The change in left prefrontal deoxygenated hemoglobin between standing and dual task walking | Baseline, within three days of completing initial open-label tDCS intervention, Month 3, Month 6, & Month 9.
  This metric is measured using functional near-infrared spectroscopy (fNIRS) and reflects one aspect of brain activation induced by performing the task of dual task walking and preferred speed.
The change in left prefrontal deoxygenated hemoglobin between standing and usual walking | Baseline, within three days of completing initial open-label tDCS intervention, Month 3, Month 6, & Month 9.
  This metric is measured using functional near-infrared spectroscopy (fNIRS) and reflects one aspect of brain activation induced by performing the task of usual walking and preferred speed.
Left dorsolateral prefrontal cortex (dlPFC) gray matter volume | Baseline & Month 3
  This metric quantifies the volume of gray matter within the left dorsolateral prefrontal cortex (the brain target-of-interest for the tDCS intervention).
Left dorsolateral prefrontal cortex (dlPFC) functional connectivity | Baseline & Month 3
  This metric quantifies the strength of functional connectivity between the left dorsolateral prefrontal cortex (the brain target-of-interest for the tDCS intervention) and the rest of the brain.
7-day accelerometry-based physical activity | Baseline, within three days of completing initial open-label tDCS intervention, Month 3, Month 6, & Month 9.
  This metric assesses the quantity and quality of habitual, real-world physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Manor, PhD, Principal Investigator — Hebrew SeniorLife; Jeff Hausdorff, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (2):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified demographic, cognitive, motor, clinical, gait kinematics, free-living accelerometry, functional near infrared spectroscopy (fNIRS), MRI, and trial compliance and safety data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Sharing of clinical trial data (participant level and summary level data, raw and processed) is expected at the time of publication of the primary results or within 9 months of database lock, whichever comes first. At minimum, per HSL's Record Management, Retention, Disposition and Destruction Policy, all data will be retained for at least seven years after project completion or the sponsored award agreement end date as stipulated in its terms and conditions.
Access Criteria: De-identified data and all metadata will be archived within the Marcus Institute Data Archiving Service (MIDAS), a publicly accessible website built on the CKAN (Comprehensive Knowledge Archive Network) open-source data management platform. The MIDAS system is maintained and hosted by Hebrew SeniorLife.
  Access to scientific data will be controlled prior to publication of the primary results or for 9 months following database lock, whichever comes first. During this period, the project PI will maintain and chair a standing subcommittee of the project investigators which will review each request. Upon majority approval of a request, access to the data may be granted in secure fashion. After this period, archived data will be accessible by investigators without need of approval by the study team. Moreover, investigators who wish to access data will not need to be affiliated with HSL. Data containing patient identifiers or related sensitive fields will be archived on HSL private servers.
URL: https://www.marcusinstituteforaging.org/